CLINICAL TRIAL: NCT06618937
Title: Toward Personalized Medicine to Guide Drug Withdrawal in Children with Juvenile Idiopathic Arthritis in Clinical Remission: a Randomized Clinical Trial Comparing Early Versus Late Drug Withdrawal Combining Imaging and Multi-Omics
Brief Title: Toward Personalized Medicine to Guide Drug Withdrawal in Children with Juvenile Idiopathic Arthritis in Clinical Remission
Acronym: Re-JIA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Nicolino Ruperto, MD, MPH, Trial Centre Director, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-514732-24-00
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
Keywords: JIA; imaging; omics; withdrawal
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biomarker-guided drug withdrawal (Experimental): Patients with inactive disease, absence of sublinical synovitis at the joint level and normal S100A8/9 and hs-CRP leves will be randomly assigned to either an early biomarker-guided drug withdrawal protocol (interventional arm) or continuation of ongoing therapy at unchanged dose for an additional 6 months and then gradual tapering (control arm).
  Patients will be evaluated at baseline, then every 3 months if still on treatment and every 6 months after drug withdrawal. At each timepoint the following procedures will be performed: joint assessment, Physician's Global Assessment of Overall Disease Activity, JAMAR, Uveitis assessment (in ANA positive patients), Hematology, chemistry, CRP, ESR, urine analysis according to drug specific schedule and Good Clinical Practice (GCP). Drug Adverse Events will be collected (MedDRA).
  MSUS and serum biomarkers quantification (S100A8/9, hs-CRP) will be repeated every 3 months until month 18 in patients with subclinical synovitis and pathologic values
  Interventions: Other: Treatment medication withdrawal strategy
- Gradual tapering (No Intervention): The control arm will continue ongoing therapy at unchanged dose for an additional 6 months and then will gradually taper the therapy.

INTERVENTIONS:
Other: Treatment medication withdrawal strategy — The study aims to compare early biomarkers-guided versus conventional unguided drugs withdrawal strategy.
  Arms: Biomarker-guided drug withdrawal

SUMMARY:
Biologic therapies made clinical remission an achievable goal for most juvenile idiopathic arthritis (JIA) patients. Nevertheless, antirheumatic drugs have side effects and are costly. Currently, no guidelines exist for withdrawing drugs in JIA patients with clinical inactive disease (CID). Relapses following the withdrawal of antirheumatic drugs are common. To establish an optimal timeline for treatment discontinuation is a major unmet need in pediatric rheumatology.

It is hypothesized that biomarkers-guided early withdrawal of antirheumatic drugs in patients achieving clinical, imaging and biological remission is safe and more effective compared to the standard practice of maintenance of stable treatment over 12 months.

DETAILED DESCRIPTION:
The study is designed as a multicenter, prospective, randomized, open label superiority trial of two different treatment medication withdrawal strategies (early biomarkers-guided versus conventional unguided drugs withdrawal strategy). Musculoskeletal ultrasound (MSUS) and serum biomarkers, such as the S-100 protein family, allow a more accurate assessment of remission status than clinical evaluation alone. Subclinical synovitis detected by MSUS at the joint level and increased level of S100 proteins have been associated with an increased risk of loss of clinically inactive disease after drug discontinuation. The results of this study will provide a more rational approach to treatment withdrawal in inactive JIA patients. It is expected that a risk-adapted strategy would reduce both number of disease flares and cumulative drug exposure compared with standard-of-care practice. If validated, these biomarkers will help to personalize immunosuppressant withdrawal: a therapy paradigm shift while ensuring patient and economic benefits.

Patients with inactive disease, absence of sublinical synovitis at the joint level and normal S100A8/9 and hs-CRP leves will be randomly assigned to either an early biomarker-guided drug withdrawal protocol (interventional arm) or continuation of ongoing therapy at unchanged dose for an additional 6 months and then gradual tapering (control arm).

Patients will be evaluated at baseline, then every 3 months if still on treatment and every 6 months after drug withdrawal. At each timepoint the following procedures will be performed: joint assessment, Physician's Global Assessment of Overall Disease Activity, JAMAR, Uveitis assessment (in ANA positive patients), Hematology, chemistry, CRP, ESR, urine analysis according to drug specific schedule and Good Clinical Practice (GCP). Drug Adverse Events will be collected (MedDRA).

MSUS and serum biomarkers quantification (S100A8/9, hs-CRP) will be repeated every 3 months until month 18 in patients with subclinical synovitis and pathologic values of serum biomarkers who are randomized in the intervention arm.

Blood samples for research laboratory analysis (multi Omics, characterization of immune cell populations and quantification of cytokines concentration and EV-miRNAs expression) will be collected at baseline, at drugs withdrawal and in case of disease flare.

ELIGIBILITY:
Inclusion Criteria:

* - Children with a diagnosis of JIA according to the ILAR classification criteria
* JIA patients who satisfy criteria for inactive disease for a minimum of 6 continuous months while still taking medication.
* Patients who have been treated with cs/b/bs/ts DMARDs according to the label indication
* Ability to comply with the entire study procedures, ability to communicate meaningfully with the investigational staff, competence to give written informed consent; to be applied to the parents and/or patients, as appropriate
* Duly executed, written, informed consent obtained from the patient's parents/legal guardian
* Female of child-bearing potential must have a negative pregnancy test at the beginning of the trial. If sexually active, they must have no intention of conceiving while on treatment with antirheumatic drugs.

Exclusion Criteria:

* - Patients with systemic JIA according to ILAR criteria
* Patients with undifferentiated arthritis according to ILAR criteria
* Patients with severe disease-related ocular damage and who need systemic treatment for uveitis
* Patients who received glucocorticoid treatment 3 months prior to baseline visit
* Patients who had previously unsuccessfully attempted tapering cs/b/bs/tsDMARDs
* Patients with severe damage as per caring physician measured
* Prior or current history of other significant concomitant illness(es) that, according to the Investigator's judgment, would adversely affect the patient's participation in the study
* Any other medical condition or laboratory examination which in the opinion of the caring physician should exclude the patient from participation to the study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of early biomarker-guided withdrawal of antirheumatic agents | 12 months
  At each timepoint the following procedures will be performed: joint assessment, Physician's Global Assessment of Overall Disease Activity, JAMAR, Uveitis assessment (in ANA positive patients), Hematology, chemistry, CRP, ESR, urine analysis according to drug specific schedule and Good Clinical Practice (GCP). Drug Adverse Events will be collected (MedDRA), to measure safety and efficacy of early biomarker-guided withdrawal of antirheumatic agents in JIA patients achieving 6 months clinical inactive disease (CID) who do not have subclinical inflammation when compared to the standard practice of maintenance of stable treatment intensity over 12 months.

SECONDARY OUTCOMES:
Rate of flare | 24 months
  To compare rate and time to flare in the randomized arms. Disease flare is defined as any patient who will loose the status of inactive disease or has a clinical Juvenile Arthritis Disease Activity Score (cJADAS)10 >1.5 or 2.5 for oligoarticular or polyarticular disease, respectively and prompt the caring physician to make a major therapeutic intervention that could include an intrarticular glucocorticoid injection, the start of systemic glucocorticoid therapy, the restart of cs/b/ts-DMARDs at the conventional regimen.
  Frequencies of flares will be analyzed in both study arms and will be compared by means of the Chi-square test or the Fisher's exact test whenever appropriate. Bionomial exact 95% confidence interval will be also computed and reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Giannina Gaslini, Genoa, GE, Italy

IPD SHARING:
Plan to Share IPD: No